CLINICAL TRIAL: NCT00065364
Title: Neurodevelopment and Experience: Behavior, Quantitative EEG and MRI
Brief Title: Improving Brain Development in Medically Healthy Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD038261 (NIH)
Record Dates: First submitted 2003-07-21; First posted 2003-07-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Premature Birth
Keywords: Preterm infant; Premature infant; Developmental care; MRI; qEEG; Neurodevelopment; Behavior; Infants; NICU
MeSH Terms: conditions — Premature Birth; Behavior

INTERVENTIONS:
Behavioral: Newborn Individualized Developmental Care Assessment Program

SUMMARY:
Premature infants born between 28 and 33 weeks' gestation often have significant brain damage. Brain damage can be caused by the much greater stimulation the infant receives in the neonatal intensive care unit (NICU) as compared to the mother's womb. This study will test the effectiveness of specialized and individualized NICU developmental care in preventing brain damage.

DETAILED DESCRIPTION:
From 28 to 33 weeks' gestation, significant neurological reorganization takes place, initiating fetal behavioral individuality and capacity for extrauterine survival. Infants born at this transitional stage exhibit unexpectedly significant brain dysfunction as they develop and age. The majority of these infants will develop psychomotor, cognitive, and attentional function deficits as well as emotional vulnerability and substandard school performance. Research suggests that these symptoms are due to a central deficit in frontal lobe processing of complex information. This central deficit may result from increased vulnerability of cerebral white matter during the last trimester of gestation, its phase of most rapid development. Persistent stress due to inappropriate sensory stimulation may contribute to alteration of early brain structure and function. This study will identify specific adaptations of the preterm brain to the transient NICU experience in order to estimate the potential of such experience in remodeling neuroanatomical structure and neurodevelopmental function. Further, the study will evaluate a program of specialized developmental care within the NICU environment.

The study's specialized developmental care model views the preterm infant as a fetus and attempts to reduce the discrepancy between the technological hospital environment and the mother's womb. A developmental specialist team will support the NICU caregivers. The developmental specialists will observe the infant's behavior and use these observations to formulate descriptive neurobehavioral reports and suggestions, to structure caregiving procedures in coordination with the infant's sleep/wake cycle, and to maintain the infant's well-regulated behavioral balance. The goal of the intervention is to promote the infant's strengths while reducing the infant's self-regulatory vulnerability.

Sixty medically healthy infants born between 28 and 33 weeks' gestation will be randomly assigned to standard NICU care or specialized developmental care. Preterm infants will be compared to 30 healthy full term infants. All infants will be assessed at 42 weeks' postconceptional age in three neurodevelopmental domains: neurobehavioral function, neuroelectrophysiological function, and neuroanatomic structure. Assessments will focus on distinct regions of the brain (occipital and frontal lobes) and the corpus callosum (which connects the right and left sides of the brain).

ELIGIBILITY:
Inclusion Criteria for Preterm Infants

* Born at Brigham and Women's Hospital (BWH), Boston
* Family residence in the greater Boston area
* Gestational age at birth of 28 to 33 weeks assessed by mother's dates, the Ballard assessment, and prenatal ultrasound as available
* Birthweight, height, and head circumference appropriate (10th to 90th percentile) for gestational age
* 1 and 5 minute Apgar >= 7
* Endotracheal intubation and mechanical ventilator support, including continuous positive airway pressure (CPAP), for < 48 hours after delivery
* Normal cranial ultrasound(s) within first 7 days of life
* Mother between 15 and 39 years old
* Telephone access
* Sufficient English language facility to assure successful communication and follow-up

Exclusion Criteria for Preterm Infants

* Use of dopamine or hydrocortisone
* Chromosomal or congenital abnormalities (e.g., Down's, Turner's, Klinefelter's syndromes)
* Congenital or acquired infections (e.g., TORCH, HIV, sepsis)
* Major maternal illness; diagnosed mental and/or emotional impairment; reported alcohol, nicotine, or illegal drug use and/or positive urine toxicity screen; or chronic medication treatment (e.g., synthroid, insulin, steroids)

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90
Dates: Start 2000-05

PRIMARY OUTCOMES:
neurodevelopmental function
EEG
MRI

CONTACTS AND LOCATIONS:
Overall Officials: Heidelise Als, PhD, Principal Investigator — Harvard University
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237
- [Background] Rivkin MJ, Wolraich D, Als H, McAnulty G, Butler S, Conneman N, Fischer C, Vajapeyam S, Robertson RL, Mulkern RV. Prolonged T*2 values in newborn versus adult brain: Implications for fMRI studies of newborns. Magn Reson Med. 2004 Jun;51(6):1287-91. doi: 10.1002/mrm.20098. PMID 15170852